CLINICAL TRIAL: NCT00249080
Title: High Field MRI of Brain Iron in Neurodegenerative Disease
Brief Title: Magnetic Resonance Imaging (MRI) of Brain Iron in Neurodegenerative Disease
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: John Schenck, MD PhD; Principal Investigator, Albany Medical College
Other Study IDs: AMC-IRB-1599; A-13214
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2009-08-24 (Estimated); Status verified 2009-08

CONDITIONS: Neurodegenerative Diseases; Mild Cognitive Impairment
Keywords: 3T MRI; neurodegenerative disease; Alzheimer's disease; spectroscopy; Normal, healthy subject without memory complaint; Not pregnant; MR compatible
MeSH Terms: conditions — Neurodegenerative Diseases; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Neurodegenerative diseases, such as Alzheimer's disease, Parkinson's disease, and multiple sclerosis are recognized as a major health concern at the present time. There is information in magnetic resonance imaging (MRI) studies regarding the role of brain iron in normal brain aging that may be enhanced with the use of better scanning equipment and procedures, and by correlating this information with clinical data. This research study aims to develop and evaluate a number of techniques that can potentially improve the effectiveness of three tesla (3T) magnetic resonance imaging of neurodegenerative brain disorders.

DETAILED DESCRIPTION:
Eligibility: A healthy person without memory complaints or someone with neurodegenerative disease. However, the person should not have metal in the body (ie, pacemaker, implants, shrapnel, etc.), should not be pregnant, and should not have claustrophobic anxieties.

Study Procedures: During a regular office visit, a neurologist will perform a routine physical and neurological examination, including your medical and family history, to determine your eligibility for this study. You will then be scheduled for a series of neuropsychological tests, which take between 1 to 1.5 hours, and an MRI scan, which takes approximately 1 hour to complete. This is a longitudinal study and you may be asked to repeat these procedures approximately every six months for the duration of this 2 year project.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Healthy person without memory complaints OR person diagnosed with a neurodegenerative disease (ie, Alzheimer's disease, Parkinson's disease, multiple sclerosis)

Exclusion Criteria:

* MR contraindication such as metal in body (ie, pacemaker, implant, shrapnel, etc.)
* Pregnant
* Claustrophobic anxieties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately equal numbers of subjects with clinically diagnosed Alzheimer's disease, multiple sclerosis, Parkinson's disease and normal controls (age and gender matched).
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2005-06; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Earl A Zimmerman, MD, Study Director — Albany Medical College; John F Schenck, MD, PhD, Principal Investigator — GE Global Research Center & Neurosciences Advanced Imaging Research Center

REFERENCES:
- [Background] Schenck JF, Zimmerman EA. High-field magnetic resonance imaging of brain iron: birth of a biomarker? NMR Biomed. 2004 Nov;17(7):433-45. doi: 10.1002/nbm.922. PMID 15523705
- [Background] Schenck JF. Magnetic resonance imaging of brain iron. J Neurol Sci. 2003 Mar 15;207(1-2):99-102. doi: 10.1016/s0022-510x(02)00431-8. No abstract available. PMID 12614939
- [Background] Schenck JF. Safety of strong, static magnetic fields. J Magn Reson Imaging. 2000 Jul;12(1):2-19. doi: 10.1002/1522-2586(200007)12:13.0.co;2-v. PMID 10931560